CLINICAL TRIAL: NCT05713968
Title: Using High Resolution Impedance Manometry and Videofluoroscopic Measurements of Swallowing Function in Patients Undergoing Cervical Spine Patients
Brief Title: Swallowing Evaluation by HRIM in Patients With Cervical Spondylosis
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202211062DIND
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Upper Esophageal Sphincter Relaxing Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with EAT-10 higher than 3 or frailty questionnaire higher than 2: patients may have high risk of aspiration
  Interventions: Other: patients with EAT-10 higher than 3 or frailty questionnaire higher than 2 examined by HRIM
- patients with EAT-10 lower than 3 or frailty questionnaire lower than 2: patients may have low risk of aspiration
  Interventions: Other: patients with EAT-10 lower than 3 or frailty questionnaire lower than 2

INTERVENTIONS:
Other: patients with EAT-10 higher than 3 or frailty questionnaire higher than 2 examined by HRIM — patients with EAT-10 higher than 3 or frailty questionnaire higher than 2 examined by HRIM
  Groups: patients with EAT-10 higher than 3 or frailty questionnaire higher than 2
Other: patients with EAT-10 lower than 3 or frailty questionnaire lower than 2 — patients with EAT-10 lower than 3 or frailty questionnaire lower than 2 examined by HRIM
  Groups: patients with EAT-10 lower than 3 or frailty questionnaire lower than 2

SUMMARY:
patients with cervical spondylolysis may have swallowing or eating difficulty. In this study, we will use high resolution impedance manometry to evaluate these patients' detailed swallowing mechanisms.

DETAILED DESCRIPTION:
This study will aim to evaluate swallowing function in patients with cervical spondylolysis by using high resolution impedance manometry (HRIM) along with oral frailty and dysphagia questionnaires. Researchers will plan to enroll 50 patients to investigate this issue. The inclusion criteria will be as following:1) age higher or equal to 20 years old; 2) patients with cervical spondylolysis or associated symptoms. The exclusion criteria will be as following: major organ dysfunction, including chronic kidney disease, bleeding tendency. The primary outcome will be the upper esophageal sphincter relaxing pressure. The researchers will hope to find the swallowing dysfunction mechanisms in these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with cervical spondylosis associated symptoms or expected to undergo cervical spine surgery
* patients with associated swallowing difficulty symptoms

Exclusion Criteria:

* major organ dysfunction, such as renal insufficiency or bleeding tendency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cervical spondylolysis patients with swallowing difficulty feelings could attend this study. The researchers will hope to help these patients to find the dysphagia mechanisms. If they have to receive early swallowing rehabilitation, we could transfer them and give the rehabilitation physicians advices.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-27 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
upper esophageal sphincter pressure | 30 minutes
  upper esophageal sphincter opening ability questionnaire

IPD SHARING:
Plan to Share IPD: No
ethical issue